CLINICAL TRIAL: NCT07259239
Title: SINGapore SoniCracker IntraVascular Lithotripsy (SING IVL) Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart Centre Singapore (Other)
Collaborators: Biosensor Interventional Technologies Pte Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0308
Record Dates: First submitted 2025-10-01; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Diseases
Keywords: SING-IVL
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Equipment and Supplies

STUDY DESIGN:
Intervention Model Description: At baseline, enrolled participants will be treated with the study device - SoniCracker Intravascular Lithotripsy Balloon during routine percutaneous coronary intervention (PCI). This device consists of a single-use, sterile catheter with multiple emitters mounted on a coronary balloon. The balloon is inserted into the coronary arteries. The emitters on the balloon then create shockwaves that cause cracks the calcium of the coronary arteries. The catheter is removed after the procedure. The rest of the PCI will be performed as per regular care.
  At 30 days post PCI procedure, participants will be followed up via telephone calls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SoniCracker IVL (Experimental)
  Interventions: Device: Medical device

INTERVENTIONS:
Device: Medical device — The SoniCracker IVL is a rapid-exchange catheter with an effective length of 1420mm, with two radiopaque markers at the distal end and is coated with a hydrophilic coating from the distal tip to the wire exchange port to facilitate tracking and catheter delivery during use. The catheter lumen consists of a wire lumen, an inflation lumen, and two shockwave electrodes. The wire lumen allows passage of a 0.014" guidewire to guide the catheter into and through the lesion. The inflation lumen is filled with a 50%/50% mixture of physiological saline and contrast media to inflate and deflate the balloon. The electrode traverses the entire effective length of the catheter for lithotripsy treatment. The proximal end of the catheter features a hub with two ports, one for inflation/deflation of the balloon, and the other for connecting the electrode wires to the Coronary intravascular lithotripsy therapy device.

SUMMARY:
Interventional cardiologists are facing an increasing burden of calcified coronary arteries in keeping with an ageing population and rising prevalence of diabetes mellitus and chronic kidney disease. Heavily calcified plaques impede balloon dilatation and successful stent delivery, resulting stent under-expansion, malposition, and damage to the drug-eluting polymer coats. This translates to poorer procedural outcomes and increased risk of Major Adverse Cardiovascular Events (MACE). The investigators' proposal seeks to determine the feasibility of the SoniCracker IVL in patients with calcified coronary lesions.

DETAILED DESCRIPTION:
Coronary calcifications are one of the strongest predictors of adverse intraprocedural and long-term PCI outcomes. We believe SoniCraker IVL provides a safer and less aggressive method of calcium modification as opposed to traditional coronary atherectomy, hence translating into better clinical outcomes for patient. Although there is a commercially available IVL (Shockwave balloon) available, it is currently priced at ~ SGD 4000. The SoniCracker IVL is potentially a more cost-effective alternative to the Shockwave IVL.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at age ≥ 21 years old.
2. Patients undergoing elective/ planned PCI with at least moderate coronary calcification on angiography at the target lesion are eligible for enrolment. Moderate coronary calcification is defined as densities on only one side of the arterial wall prior to contrast injection. Severe calcification was defined as radiopacities on both sides of the arterial wall prior to contrast injection.
3. Patients need to demonstrate evidence of either a 180 arc of coronary calcium or nodular calcium at the target lesion on intravascular imaging prior to IVL therapy.

Exclusion Criteria:

1. Significant co-morbidities:

   * Cardiac arrest
   * Cardiogenic shock
   * Collapse / comatose / semi-conscious states
2. Patients requiring urgent or emergent PCI.
3. Patients who are unable to provide consent.
4. Patients who are pregnant.
5. Breast-feeding women
6. Any patients whom the Investigator deems unsuitable for the study (e.g., due to other medical reasons, laboratory abnormalities, expected study medication noncompliance, or subject's unwillingness to comply with all study-related study procedures).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Procedural success | Perioperative
  Successful delivery and deployment of the study device, and attainment of less than 50% diameter stenosis after stenting with no evidence of in-hospital major adverse cardiac events (MACE: cardiac death, myocardial infarction or target vessel revascularization)

SECONDARY OUTCOMES:
Device success (successful delivery and deployment of a device, and attainment of less than 50% diameter stenosis), 30-day MACE, coronary complications, post procedural angiographic and intravascular imaging outcomes | Up to 30 days (+ 1 month) post PCI

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart Center Singapore, Singapore, Singapore